CLINICAL TRIAL: NCT01240668
Title: An Observational Prospective Registry to Identify Demographic and Clinical Characteristics of Patients Hospitalized With Euvolemic and Hypervolemic Hyponatremia and Assess the Comparative Effectiveness of Available Treatments and the Impact on Resource Utilization
Brief Title: Hyponatremia Registry for Patients With Euvolemic and Hypervolemic Hyponatremia
Acronym: HN Registry
Status: Completed | Type: Observational
Sponsor: Otsuka America Pharmaceutical (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Other Study IDs: 156-10-292
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Euvolemic Hyponatremia; Hypervolemic Hyponatremia
Keywords: Hyponatremia; Euvolemia; Hypervolemia; Euvolemic; Hypervolemic
MeSH Terms: conditions — Hyponatremia; Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hyponatremia Patients: Euvolemic or hypervolemic hyponatremia with serum sodium ≤130 mmol/L

SUMMARY:
The registry is a multi-center, prospective, observational study designed to collect data in patients with euvolemic and hypervolemic hyponatremia in the hospital setting in the USA and hyponatremia secondary to syndrome of inappropriate antidiuretic hormone secretion (SIADH) in Europe; patients with hypovolemic hyponatremia will be excluded from the registry. The registry is observational in design, and the registry will collect data on patients with a serum sodium ≤130 mmol/L. Data from the patients' chart will be collected throughout the duration of the hospital, from admission to discharge, and the data will be entered into the case report form (CRF) or into an electronic data capture (EDC) system. These patients will be entered into the registry over the duration of 18 months at community, tertiary, and academic medical centers from diverse multiple regions of the USA and Europe.

A patient's treatment will be determined by their caregiver and not by this protocol. Thus, the registry will provide a unique opportunity to evaluate how the patients are managed under real-world management conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old who are hospitalized
* Euvolemic or hypervolemic hyponatremia with serum sodium ≤130mmol/L
* For euvolemic hyponatremia:

  * Euvolemia is defined as: absence of clinical and historical evidence of extracellular fluid volume depletion or sequestration; and absence of edema and ascites; or
  * Physician diagnosis of SIADH
* For hypervolemic hyponatremia (applies to USA sites only):

  * Hypervolemia is defined as: excess extracellular fluid volume manifesting as dependent edema or ascites
  * Patients may have one or more of the following underlying co-morbid conditions:

    * Congestive heart failure
    * Cirrhosis and/or liver failure
    * Nephrotic syndrome

Exclusion Criteria:

* Patients with hypovolemic hyponatremia
* Use of investigational drug, biologic, or device during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective registry study population will consist of up to 1500 patients at approximately 150 sites from the USA who are hospitalized and identified as having hypervolemic or euvolemic hyponatremia with serum sodium ≤130 mmol/L. Also up to 1005 patients at approximately 67 sites from Europe (United Kingdom, Germany, France, Italy, Spain, Denmark, and Sweden)who are identified as having hyponatremia ≤130mmol/L secondary to SIADH. A similar distribution of patients with a serum sodium <125 mmol/L and patients with a serum sodium between 125-130 mmol/L will be collected.
Sampling Method: Probability Sample
Enrollment: 5028 (Actual)
Dates: Start 2010-09; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in serum sodium concentration from beginning of treatment period to the end of treatment period or discharge for a given hyponatremia treatment | Hospital Discharge
Duration of hospital stay from time of first presentation of hyponatremia (which will be taken as the time of first presentation of hyponatremia for the current admission) to discharge | Hospital Discharge
Time to initiation of hyponatremia treatment | Hospital Discharge

SECONDARY OUTCOMES:
Relative proportions of etiologies associated with hyponatremia | Hospital Discharge
Profile of investigations performed in diagnosing hyponatremia | Hospital Discharge
Therapies used in the management of hyponatremia | Hospital Discharge
Effectiveness of individual therapies in correcting hyponatremia and time taken to achieve the correction. | Hospital Discharge
  Effectiveness of individual therapies in correcting hyponatremia and time taken to achieve the correction measured as one of the following:
  serum sodium >130 serum sodium ≥135 mmol/L increase of serum sodium ≥5 mmol/L
Effectiveness of individual therapies in correcting hyponatremia and time taken to achieve the correction. | Hospital Discharge
  Effectiveness of individual therapies in correcting hyponatremia and time taken to achieve the correction measured as one of the following:
  * serum sodium >130
  * serum sodium ≥135 mmol/L
  * increase of serum sodium ≥5 mmol/L
Effectiveness of individual therapies in achieving symptom improvement measured as the number of reported symptoms at the start and end of treatment with a specific therapy | Hospital Discharge
Medically necessary length of hospital stay and duration of intensive care unit (ICU) stay | Hospital Discharge
Impact of hyponatremia on medically necessary length of stay | Hospital Discharge

CONTACTS AND LOCATIONS:
Locations (79):
- United States (72):
  - North America Research Institute, Azusa, California
  - Chrishard Medical Group, Inglewood, California
  - UCLA, Los Angeles, California
  - Regional Cardiology Associates, Sacramento, California
  - Portercare Adventist Health System, Denver, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Memorial Healthcare System, Hollywood, Florida
  - Jacksonville Cardiovascular Center, Jacksonville, Florida
  - Kidney & HTN Specialists of Miami, Miami, Florida
  - Naples Community Hospital, Naples, Florida
  - Florida Hospital, Orlando, Florida
  - Coastal Nephrology Associates Research, Port Charlotte, Florida
  - St. Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Joseph M Still Research Foundation, Inc, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Research Integrity, LLC, Owensboro, Kentucky
  - Ochsner Multi-Organ Transplant Center, New Orleans, Louisiana
  - Detroit Medical Center, Detroit, Michigan
  - Detroit Receiving Hospital, Detroit, Michigan
  - Central Michigan Community Hospital, Mount Pleasant, Michigan
  - Providence Park Hospital, Novi, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Covenant Heart Specialists, Saginaw, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Saint Louis University Hosptial, St Louis, Missouri
  - Creighton University, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hypertenstion and Renal Group, Livingston, New Jersey
  - St Joseph's Regional Medical Center, Paterson, New Jersey
  - Princeton Hypertension Nephrology Associates, Princeton Junction, New Jersey
  - Tufts New England Medical Center, Boston, New York
  - Buffalo General Hospital, Buffalo, New York
  - The Jamaica Hospital Medical Center, Jamaica, New York
  - Winthrop-University Hospital, Mineola, New York
  - Beth Israel Medical Center-Petrie Division, New York, New York
  - Center for Liver Disease and Transplantation, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - NYU, New York, New York
  - Rochester General, Rochester, New York
  - University of Rochester, Rochester, New York
  - St Catherine of Siena Medical Center, Smithtown, New York
  - Jack D. Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Piedmont Respiratory Research, Greensboro, North Carolina
  - Mercy Hospital, Canton, Ohio
  - University of Cinncinati, Cincinnati, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Mercy Hospital Fairfield, Fairfield, Ohio
  - Kettering Health Network, Kettering, Ohio
  - Kidney Care Specialists, Kettering, Ohio
  - St Elizabeth Health Center, Youngstown, Ohio
  - NE Clinical Research Center, Bethlehem, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Heart Specialists of Lancaster PC, Eprata, Pennsylvania
  - Laurel Health System, Mansfield, Pennsylvania
  - UPMC Center for Liver Disease, Pittsburgh, Pennsylvania
  - SC Nephrology & Hypertension Ctr, Orangeburg, South Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Saint Thomas Hospital, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Cardiopulmonary Research Science & Technology Institute, Dallas, Texas
  - Baptist Hospital Downtown, San Antonio, Texas
  - Renal Associates, PA, San Antonio, Texas
  - Clinical Research and Consulting Centter, Fairfax, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - CAMC Institute Inc., Charleston, West Virginia
- Germany (4):
  - Evangelische Lungenklinik, Berlin
  - Klinikum Chemnitz, Chemnitz
  - Universitätsklinik Köln, Cologne
  - Klinikum der Johann-Wolfgang-Goethe-Universität, Frankfurt
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Liverpool University Hospital, Liverpool
  - Royal Victoria Infirmary, Newcastle